CLINICAL TRIAL: NCT05465824
Title: Risk Stratification of Patients With Suspected COVID-19 Presenting to the ED
Acronym: EuroCOV
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Principal Investigator, Saïd LARIBI, Principal Investigator, University Hospital, Tours
Other Study IDs: EuroCOV
Record Dates: First submitted 2022-03-10; First posted 2022-07-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive study of patients with suspected COVID-19 upon ED arrival of European hospitals between March 09 and April 08 2020.

Justification:

DETAILED DESCRIPTION:
Descriptive study of patients with suspected COVID-19 upon ED arrival of European hospitals between March 09 and April 08 2020.

Justification:

Over the past 3 months, the world has faced a novel infection disease outbreak, due to a novel coronavirus, the severe acute respiratory syndrome coronavirus (SARS-CoV2), with a massive impact on healthcare resource.

In Europe, numbers of confirmed cases continue to rise. Europe is currently one of the regions with the highest number of Covid-19 cases and deaths due to this emergent diseases.

Most COVID-19 infected patients present with mild to moderate acute respiratory symptoms, including cough, fever, dyspnea and pneumonia. About 20% will present with severe or critical manifestations of the disease, including pneumonia, respiratory failure and acute respiratory distress syndrome (ARDS).

Anticipating the needs for hospitalization in ward and/or intensive care is crucial.

Emergency departments are at the front line for triaging patients with suspected Covid-19 and referring them to the appropriate level of care.

In Europe, the number of ED patients with suspected Covid-19 is variable; rate of hospitalization from ED reaches 40% for this population.

Risk stratification and management decisions of patients presenting to the ED with suspected COVID-19 is a challenge for emergency physicians.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (>= 18 years old) attending the ED with a clinical suspicion of COVID-19 based on the presence of the following criteria

* Fever >= 38 °C
* respiratory symptoms (dyspnea, cough, expectorations)
* any other symptoms suggestive of COVID-19 including digestive signs (diarrhea, anosmia…)

Exclusion Criteria:

* No insurance
* patients less than 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a suspected Covid 19
Sampling Method: Non-Probability Sample
Enrollment: 7876 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 30 days
  Mortality during hospital management

CONTACTS AND LOCATIONS:
Locations (1):
- Tours University Hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided